CLINICAL TRIAL: NCT04930588
Title: Gingival Crevicular Fluid and Salivary Levels of Neuregulin-4 and Its Receptor ErbB4 in Patients With Stage III and IV Periodontitis With and Without Type 2 Diabetes: An Observational Study
Brief Title: Levels of Neuregulin-4 and Its Receptor ErbB4 in Periodontitis Patients With and Without Diabetes Type 2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Samir Abdel Fatah, Asmaa Samir, Cairo University
Other Study IDs: PER7-2-1
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Periodontitis; Diabetes Mellitus
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to assess the levels of neuregulin-4 and its receptor ErbB4 in the GCF and saliva in stage III and IV periodontitis patients with and without type 2 diabetes mellitus.

DETAILED DESCRIPTION:
The aim of this study is to measure the levels of Nrg4 and ErbB4 in the GCF and saliva of periodontitis stage III and IV patients with and without type 2 diabetes mellitus and to correlate their levels with the periodontal clinical parameters and the blood glucose levels including the fasting plasma glucose level (FPG) and glycated hemoglobin (HbA1c).

This study will be conducted in the Oral Medicine and Periodontology department, Faculty of Dentistry- Cairo University, Egypt.

Patients will be selected from the outpatient clinic of the department of Oral Medicine and Periodontology, Faculty of Dentistry-Cairo University.

ELIGIBILITY:
Inclusion Criteria:

* For periodontitis stage III and IV patients according to (Papapanou et al., 2018 and Tonetti et al., 2018)

  1. Bleeding on probing (BOP) ≥ 30%.
  2. At least four non-adjacent teeth sites in each jaw having CAL ≥ 5 mm and PD ≥ 6 mm in one or more sites.
  3. Tooth loss due to periodontitis ≥ 5 teeth.
  4. Presence of a minimum of 15 natural teeth. For diabetes and non-diabetic patients according to ("Diagnosis and Classification of Diabetes Mellitus," 2014)
  5. Patients with type 2 diabetes mellitus will be diagnosed as having type 2 diabetes mellitus ≥ 5 years before the study and treated with stable doses of oral hypoglycaemic agents and/or insulin under the supervision of an endocrinologist with their glycated haemoglobin level (HBA1c) > 6%.
  6. Non diabetic Patients in the control and stage III and IV periodontitis groups will be selected as having Fasting plasma glucose (FPG) <126 mg/dL.

Exclusion Criteria:

1. Individuals with any known systemic disease other than type 2 diabetes.
2. Pregnant and lactating women.
3. Individuals that received periodontal treatment within the last 6 months.
4. Individuals with a history of systemic antibiotics and anti-inflammatory drugs within the last 3 months.
5. Former or current smokers.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Dental patients will be recruited in a consecutive manner from the clinic of the department of Oral Medicine and Periodontology, Faculty of Dentistry -Cairo University.
  Medical history and dental history will be taken; thorough oral examination will be done.
  The aim of the study will be explained to the patient and the patient's acceptance to participate in the survey will be received.
  Non-respondent patients or patients refusing to participate will be reported with the cause of their refusal.
  Conventional oral and periodontal examination will be held on a dental unit using the light of the unit, mirror and probe
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Neuregulin-4 in the GCF | 6 month
  Measured by Enzyme-Linked Immunosorbent Assay in μL
The receptor ErbB4 in the GCF | 6 month
  Measured by Enzyme-Linked Immunosorbent Assay in μL
Neuregulin-4 in the saliva | 6 month
  Measured by Enzyme-Linked Immunosorbent Assay in μL
The receptor ErbB4 in saliva | 6 month
  Measured by Enzyme-Linked Immunosorbent Assay in μL

SECONDARY OUTCOMES:
Pocket depth | 6 month
  Measured by Manual UNC periodontal probe in mm
Clinical attachment level | 6 month
  Measured by Manual UNC periodontal probe in mm
Bleeding on probing | 6 month
  Measured by Manual UNC periodontal probe by gently probing the orifice of the gingival crevice, the periodontal probe will be inserted 1 to2 mm into the gingival sulcus starting at one interproximal area and moving to the other. If bleeding occurs within 10 seconds a positive finding is recorded.
plaque index | 6 month
  Measured by Manual UNC periodontal probe Scores:
  0: No plaque
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of a disclosing solution or by using the probe on the tooth surface.
  2. Moderate accumulation of soft deposits within the gingival pocket, or the tooth and gingival margin, which can be seen with the naked eye.
  3. Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Glycosylated Haemoglobin (HbA1c %) | 6 month
  Measured by High performance liquid chromatography in mmol/mol
Fasting plasma Glucose Level (FPG) | 6 month
  Measured by blood sampling in (mg/dl)
Body Mass Index (BMI) | 6 month
  Measured in (Kg/m2)

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa samir, master, Principal Investigator — Cairo University
Locations (1):
- Cairo university Faculty of dentistry, Cairo, Egypt